CLINICAL TRIAL: NCT07017153
Title: Evaluation of the Impact of Decision Aids on Treatment Choices in Patients With Arterial Hypertension: A Pilot Study
Brief Title: Patient Decision Aids for Hypertension: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medizinische Hochschule Brandenburg Theodor Fontane (Other)
Responsible Party: Principal Investigator, Jan Berghold, Medical Student and Doctoral Candidate, Medizinische Hochschule Brandenburg Theodor Fontane
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 260112024-ANF
Record Dates: First submitted 2025-04-16; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Patient Decision Aid
Keywords: arterial hypertension; patient decision aid; shared decision making; decision aid; patient engagement; pilot study; adherence
MeSH Terms: conditions — Hypertension; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient Decision Aid B (Other): Patients will receive Decision Aid B. Original:
  "How Do I Control My Blood Pressure? Lifestyle Options and Choices of Medicines". (NICE 2019. ISBN 978-1-4731-3543-7) German Translation for our Study: "Wie kann ich meinen Bluthochdruck behandeln? Optionen zu Lebensstiländerungen und der Medikamentenwahl"
  Interventions: Other: Questionnaire B
- Patient Decision Aid A (Other): Patients will receive Decision Aid A. Original: "Bluthochdruck - Wie Herz-Kreislauf-Erkrankungen vorbeugen?". (SHARE TO CARE, 2025. https://entscheidungshilfe.share-to-care.de/bluthochdruck/ (access: 25.02.2025)) English translation: "Hypertension - How to Prevent Cardiovascular Diseases"
  Interventions: Other: Questionnaire A

INTERVENTIONS:
Other: Questionnaire B — Questionnaire regarding patient decision aid: How Do I Control My Blood Pressure? Lifestyle Options and Choices of Medicines.
  Arms: Patient Decision Aid B
Other: Questionnaire A — Questionnaire regarding patient decision aid: Hypertension - How to Prevent Cardiovascular Diseases
  Arms: Patient Decision Aid A

SUMMARY:
Background: Arterial hypertension is a major global health problem with a leading cause of premature death and a major risk factor for cardiovascular disease. Despite its prevalence, blood pressure control remains suboptimal, requiring effective treatment and patient engagement strategies. With the increasing emphasis on person-centered care, healthcare professionals and patients are moving toward shared decision-making (SDM), which is defined as an approach to collaboratively making health decisions in line with recent evidence and patient preferences and values. Patient decision aids (PDAs) are tools designed to involve patients in treatment decisions by providing clear information about options, benefits and risks, while helping them to clarify personal values. These tools have been shown to improve decision quality, adherence and health outcomes.

Methods: This pilot study aims to evaluate the practical utility of two PDAs with different formats for antihypertensive therapy from the patient's perspective. Adult patients (≥ 18 years) with hypertension admitted to a university hospital will be randomized to use one of the two PDAs displayed on a tablet. After viewing the PDA, participants will complete a questionnaire assessing their knowledge, risk perception, preferences, and involvement in decision-making. Descriptive statistics will be used to analyze the data.

Expected results: The study anticipates that the PDAs will increase patients knowledge of treatment options, support value clarification and improve engagement in SDM. These findings will inform the design of a larger randomized controlled trial to optimize PDA formats for hypertension management.

DETAILED DESCRIPTION:
Detailed Description

1. INTRODUCTION Arterial hypertension is one of the most important modifiable risk factors for cardiovascular disease and a leading cause of premature death worldwide. Despite effective therapies, only about 20% of the 1.28 billion adults worldwide have their blood pressure under control, increasing the risk of major cardiovascular events. This highlights the need for personalized treatment strategies and patient engagement. Shared decision-making (SDM) is a key approach to collaborative decision-making between patients and healthcare professionals, aimed at tailoring treatment options and goals to patients' needs and preferences, as emphasized in the ESC 2024 guidelines. Patient decision aids (PDAs) are tools designed to support SDM by providing clear information about treatment options, risks and benefits, while helping patients to clarify their preferences and values. Evidence suggests that PDAs improve the quality of decisions, promote adherence and have a positive impact on hypertension outcomes.
2. BACKGROUND AND RATIONALE Hypertension management requires a patient-centered approach, as treatment goals, such as achieving a target systolic blood pressure of 120-129 mmHg, should be adapted to individual tolerance and well-being. The 2024 ESC guidelines highlight the importance of SDM. PDAs can help overcome challenges. These tools prepare patients to make value-based decisions without replacing medical consultations. Despite their potential benefits, there is limited evidence on which PDA format and features are most effective for hypertensive patients. This pilot study aims to address this gap by evaluating different PDA formats to identify those that best improve patient understanding, knowledge and value clarification. The results will inform the design of optimized PDAs for clinical use in hypertension management and contribute to overcoming existing barriers to SDM in practice.
3. OBJECTIVES The aim of this pilot study is to evaluate PDAs for antihypertensive therapy from the patient's perspective to answer the following research question: Which format of PDA is most useful in practice to support SDM in hypertension management?

Specifically, the study aims to:

1. Evaluate which design features of two different PDA formats are most effective improving patients knowledge of hypertension management regarding the available treatment options, including their benefits and risks.
2. Evaluate how PDAs support patients in clarifying their personal values and preferences regarding treatment choices.
3. Investigate whether the use of PDAs increases patients involvement in SDM. Findings will inform the development of optimized PDA formats that can improve patient adherence, enhance decision quality, and ultimately contribute to better clinical outcomes in hypertension care.
4. METHODS Study design: Randomized controlled pilot study to assess which format of PDAs is most useful in supporting SDM about antihypertensive therapy and to identify potential challenges and refine the methodology for a future large-scale trial. Participants: the study will include a minimum of 60 adult patients (≥ 18 years) diagnosed with arterial hypertension of any grade and regardless of the time of diagnosis. Patients need to be treated at the Department of Internal Medicine I, University Hospital Brandenburg an der Havel, Germany. Eligible participants will be invited to participate regardless of their reason for hospitalization, provided they meet the inclusion criteria. Randomization: Participants will be randomly allocated to one of two intervention arms using a computer-generated allocation sequence. Intervention arm A:

   Participants will use the decision aid "How so I control my blood pressure? Lifestyle options and choices of medicines." (https://www.nice.org.uk/guidance/ng136/resources/how-do-i-control-my-blood-pressure-lifestyle-options-and-choice-of-medicines-patient-decision-aid-pdf-6899918221) Intervention arm B: Participants will use the decision aid "Bluthochdruck - Wie Herz-Kreislauf-Erkrankungen vorbeugen?" (engl.: High Blood Pressure - How to prevent cardiovascular disease). (https://entscheidungshilfe.share-to-care.de/bluthochdruck/)

   Intervention: Participants in each arm will review their assigned PDA on a tablet computer. The two formats will be compared based on their ability to facilitate patient understanding and value clarification. Data collection: After using the assigned PDA, participants will complete a questionnaire designed to address the following aspects:
   * Knowledge of hypertension and treatment options.
   * Perceived risk of untreated or poorly controlled hypertension.
   * Patient-reported involvement in the decision-making process.
   * - Personal values and preferences influencing treatment choices (e.g. lifestyle changes, medication or combination of therapies).
   * Confidence in the decision-making process supported by the PDA.
   * Expected health outcomes and satisfaction with the usability of the PDA. Statistical Analysis: Descriptive statistics will be used to summarize participant characteristics and questionnaire responses in each intervention arm. Comparative analysis between groups will identify differences in knowledge acquisition, risk perception, value clarification, and overall satisfaction with the decision-making process supported by each of the two PDAs .
5. Timeline The pilot study is expected to be completed within 2 months (date: 30.04.2025).
6. Ethical considerations Ethical approval for this study was obtained from the Ethics Committee of the Brandenburg Medical School - Theodor Fontane prior to commencement of the study (waiver no. 260112024). Written informed consent will be obtained from all participants prior to enrolment.
7. Dissemination plan: The aim is to disseminate the study results with a focus on reaching and informing PDA developers through target journals. Target group: PDA developers, health professionals, researchers.

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years)
* Diagnosed with hypertension (all stages), regardless of primary reason for treatment.
* Receiving treatment at the Department of Internal Medicine I, University Hospital Brandenburg an der Havel

Exclusion Criteria:

* Patients under 18 years old
* Pregnancy-induced hypertension
* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Patient-perceived usefulness of hypertension decision aids | Up to 24 weeks
  Patient-Perceived Usefulness of the Decision Aid (Measured by a Study-Specific Questionnaire adapted from the Multidimensional Measure of Informed Choice [MMIC; DOI: 10.1016/S0738-3991(02)00089-7], assessing relevance, clarity, and ease of use, aligning with questions addressing decision aids for arterial hypertension therapy)

SECONDARY OUTCOMES:
Knowledge | Up to 24 weeks.
  Patient knowledge: "Patient knowledge about hypertension and treatment options (measured by a study-specific knowledge questionnaire that assesses understanding of blood pressure targets, medication side effects, and lifestyle changes, and is consistent with questions on data collected at enrolment)."
  Self-rated knowledge is assessed using a 5-point Likert scale for each item, with response options ranging from "Sehr gut" (very good, scored as 1) to "Sehr gering" (very poor, scored as 5). Thus, lower scores indicate better self-rated knowledge. The minimum score per item is 1, the maximum is 5.
  Knowledge of treatment options is assessed by a multiple-choice question with 17 possible options (including "Keine" (none)). The score is the number of correct options selected (minimum = 0, maximum = 16; higher scores indicate better knowledge of treatment options).
Risk Perception | Up to 24 Weeks
  Risk perception: "Patient perception of risk related to hypertension (measured by a study-specific risk perception scale assessing the perceived likelihood and severity of cardiovascular events, aligned with questions on data collected at enrolment)".
  Sociodemographic and health-related data are collected at enrolment: sex (male, female, no answer), date of birth (free text), height (cm) and weight (kg, free text), highest educational attainment (14 options), smoking status (never, former, occasional, regular, daily), physical activity (never, 1-2, 3-4, 5+ times/week), cholesterol (yes, no, unknown), diabetes (yes, no, unknown), and family history of premature cardiovascular events (father, mother, brother, sister, no, unknown).
Confidence in decision-making | Up to 24 Weeks
  Confidence in decision-making: "Patient confidence in making decisions about hypertension treatment (measured by a study-specific confidence scale assessing sense of control, understanding of options, and ability to weigh pros and cons, aligned with questions addressing data collected during enrolment)".
  Responses are collected using a 5-point Likert scale for each item: 1 = "Ja, auf jeden Fall"/"Ja, definitiv" (definitely yes), 2 = "Ja, wahrscheinlich"/"Eher ja" (probably yes), 3 = "Neutral", 4 = "Wahrscheinlich nicht"/"Eher nein" (probably not), 5 = "Nein, auf keinen Fall" (definitely not). The minimum score per item is 1, the maximum is 5. Lower scores indicate greater confidence or acceptance.
Preparation for decision making | Up to 24 weeks
  Preparation for decision making: "Patient preparation for decision making regarding hypertension treatment.
  This outcome is measured using a study-specific questionnaire (LimeSurvey), which includes multiple 5-point Likert scale items (e.g., perceived helpfulness, knowledge gain, support for informed decision making) as well as open-ended questions. For each Likert scale item, responses are scored from 1 (most positive, e.g., "Sehr hilfreich", "Sehr gut informiert", "Ja vollständig") to 5 (most negative, e.g., "Überhaupt nicht hilfreich", "Überhaupt nicht informiert", "Überhaupt nicht"). Minimum score per item is 1, maximum is 5; lower scores indicate greater preparation for decision making.

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Universitätsklinikum Brandenburg an der Havel, Hochstraße 29, 14770 Brandenburg an der Havel, Brandenburg, Brandenburg
  - Institute for Health Services and Health System Research, Faculty of Health Science Brandenburg, Brandenburg Medical School (Theodor Fontane), Rüdersdorf, Brandenburg

IPD SHARING:
Plan to Share IPD: No
While the results of this study will be published, including aggregated data and findings, individual patient data (IPD) will generally not be shared. We are committed to protecting the privacy of our patients. If sharing of anonymised IPD is considered in the future for collaborative research purposes, it will only be done with the explicit further consent of participants and in accordance with all applicable data protection regulations. The possibility of sharing and the conditions under which it would occur will be reassessed at that time.

REFERENCES:
- See also: Intervention Arm B: How do I control my blood pressure? Lifestyle options and choice of medicines Patient decision aid — https://www.nice.org.uk/guidance/ng136/resources/how-do-i-control-my-blood-pressure-lifestyle-options-and-choice-of-medicines-patient-decision-aid-pdf-6899918221
- See also: Intervention Arm A: Bluthochdruck - Wie Herz-Kreislauf-Erkrankungen vorbeugen? (user: Innovationsfonds_SDM pw: Making_SDM_a_Reality) — https://entscheidungshilfe.share-to-care.de/bluthochdruck/meine-erkrankung/was-bedeutet-meine-erkrankung/
- See also: World Health Organization: Hypertension — https://www.who.int/news-room/fact-sheets/detail/hypertension
- See also: International Patient Decision Aid Standards Collaboration: What are patient decision aids? — https://decisionaid.ohri.ca/IPDAS/what.html
- See also: Kim S, Shin DW, Yun JM, Hwang Y, Park SK, Ko YJ, Cho B. Medication Adherence and the Risk of Cardiovascular Mortality and Hospitalization Among Patients With Newly Prescribed Antihypertensive Medications. Hypertension. 2016 Mar;67(3):506-12. doi: 10.1161 — https://pubmed.ncbi.nlm.nih.gov/26865198/